CLINICAL TRIAL: NCT05642832
Title: Feasibility of Reducing Respiratory Drive in Patients with Acute Hypoxemic Respiratory Failure Using the Through-flow System
Brief Title: Feasibility of Reducing Respiratory Drive Using the Through-flow System
Acronym: Throughflow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-5534
Record Dates: First submitted 2022-07-14; First posted 2022-12-08 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Insufficiency; Diaphragm Injury; Lung Injury
MeSH Terms: conditions — Respiratory Insufficiency; Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Throughflow (Experimental): Throughflow is a novel system that reduces anatomical dead space by providing a constant flow of fresh gas (i.e., gas that is free of CO2) during inspiration in patients receiving invasive mechanical ventilation. By clearing the CO2 that normally remains in the upper airway after exhalation (anatomical dead space), TF can dramatically reduce anatomical dead space without the need to increase the delivered VT, making it a safe strategy in terms of lung protection. This reduction in dead space reduces the ventilatory demands of the patients, reducing respiratory drive.
  Interventions: Device: Throughflow titration phase

INTERVENTIONS:
Device: Throughflow titration phase — Ventilation will be applied in the TF mode with TF set to 0 LPM for 10 minutes. Patients will receive assist through the NAVA line of the tri-piece (NAVA set to similar settings as Servo period, ~60-80 LPM flow). Ventilation with Throughflow will be started at a TF flow of 5 LPM, and the NAVA flow will be reduced by 5 LPM. After 10 minutes measurements will be collected. If Edi is greater than or equal to 4 µV, TF flow will be increased to 10 LPM and NAVA flow will be adjusted to keep total flow constant. Measurements will be collected again after 10 minutes. TF flow will be increased in steps of 5 LPM and measurements collected every 10 minutes until Edi is below 3 µV or TF flow reaches the total flow observed during the NAVA period.
  After either the Edi target has been met or TF flow has reached the total flow, ventilation with TF will be reduced in steps of 5 LPM every 10 minutes (the reverse of the above), while NAVA flow is accordingly adjusted to keep total flow constant.

SUMMARY:
Mechanical ventilation can lead to diaphragm and lung injury. During mechanical ventilation, the diaphragm could be completely rested or it could be overworked, either of which may cause diaphragm injury. Mechanical stress and strain applied by mechanical ventilation or by the patient's own respiratory muscles can also cause injury to the lungs. Diaphragm and lung injury are associated with increased morbidity and mortality. Throughflow is a novel system that can reduce dead space without the need to increase the tidal ventilation, reducing the ventilatory demands and respiratory drive.

DETAILED DESCRIPTION:
Patients with acute respiratory failure often develop significant diaphragm weakness during mechanical ventilation. Diaphragm weakness is associated with prolonged duration of mechanical ventilation and higher risk of death. Clinical data and experimental evidence indicate that the ventilator injures the diaphragm via two opposing mechanisms, disuse and excessive loading. Cessation of diaphragm activity leads to rapid disuse atrophy within hours. On the other hand, high inspiratory loads result in myofibril edema, inflammation and contractile dysfunction. In light of this, studies found that patients with an intermediate level of inspiratory effort, similar to that of healthy subjects breathing at rest, exhibited the shortest duration of ventilation.

Arterial CO2 (PaCO2) tension and physiological dead space play an important role in determining the ventilatory requirements and respiratory drive in patients with AHRF.

Throughflow (Neurovent) is a novel system that reduces anatomical dead space by providing a constant flow of fresh gas (i.e., gas that is free of CO2) during inspiration in patients receiving invasive mechanical ventilation. By clearing the CO2 that normally remains in the upper airway after exhalation (anatomical dead space), TF can dramatically reduce anatomical dead space without the need to increase the delivered VT.

Reducing dead space offers a theoretical benefit in mitigating the mechanisms of lung and diaphragm injury during spontaneous breathing by reducing the ventilation demands to the lungs. Animal studies using the TF have shown extremely promising results, however, the impact of reducing anatomical dead space using the TF on gas exchange, ventilation, and respiratory drive in critically ill patients with AHRF is unknown.

ELIGIBILITY:
Inclusion Criteria:

* PaO2/FiO2 less than or equal to 300 at time of screening
* Oral endotracheal intubation with ETT 7.5 or 8.0 and on invasive mechanical ventilation
* Bilateral airspace opacities on chest radiograph or chest CT scan

Exclusion Criteria:

* Contraindication to esophageal catheterization (upper gastrointestinal tract surgery within preceding 6 weeks, bleeding esophageal/gastric varices)
* Intubation for traumatic brain injury or stroke
* Intracranial hypertension (suspected or diagnosed by medical team)
* Anticipated liberation from mechanical ventilation within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Esophageal pressure swing (respiratory effort) | 24 hours
  Changes in esophageal pressure swing from baseline to protocol completion will be described using central tendency and dispersion measurements (median and 25%-75% interquartile range) for each variable at each time point of the protocol
Dynamic driving transpulmonary pressure (lung-distending pressure) | 24 hours
  Changes in the dynamic driving transpulmonary pressure from baseline to protocol completion will be described using central tendency and dispersion measurements (median and 25%-75% interquartile range) for each variable at each time point of the protocol
Oxygenation (PaO2/FiO2 ratio) | 24 hours
  Changes in PaO2/FiO2 from baseline to protocol completion will be described using central tendency and dispersion measurements (median and 25%-75% interquartile range) for each variable at each time point of the protocol

SECONDARY OUTCOMES:
Rate of serious adverse events | 24 hours
  The number of SAEs during the protocol will be measured and quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto; Lorenzo Del Sorbo, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No